CLINICAL TRIAL: NCT00837096
Title: A Prospective, Randomized, Multicenter, Parallel Study Comparing V.A.C. Negative Pressure Wound Therapy (NPWT) to Moist Wound Therapy (MWT) in the Treatment of Diabetic Foot Amputation Wounds
Brief Title: A Study Comparing V.A.C. Negative Pressure Wound Therapy (NPWT) to Moist Wound Therapy (MWT) in the Treatment of Diabetic Foot Amputation Wounds
Acronym: VAC 2006-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business objectives changed.
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAC 2006-19
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Amputation Foot Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V.A.C. Therapy (Experimental): Negative Pressure Wound Therapy (NPWT) distrubtes negative pressre across a wound base by means of a specially engineered dressing with the specific intent to help promote wound healing.
  Interventions: Device: V.A.C. Therapy
- Moist Wound Therapy (MWT) (Active Comparator): t wound therapy (MWT) is a widely used treatment modality that demonstrates benefit through the facilitation of a moist wound environment, which is known to promote faster relative wound healing compared to wounds exposed to air.
  Interventions: Device: Moist wound therapy (MWT)

INTERVENTIONS:
Device: V.A.C. Therapy — Negative Pressure Wound Therapy (NPWT) distributes negative pressure across a wound base by means of a specially engineered dressing with the specific intent to help promote wound healing.
  Arms: V.A.C. Therapy
Device: Moist wound therapy (MWT) — Gauze Pads, Transparent Films, Hydrogels, Foam, Hydrocolloids, alginate, collagen, and antimicrobial
  Arms: Moist Wound Therapy (MWT)

SUMMARY:
The objective of this study is to thoroughly examine the role of V.A.C. NPWT in the further salvage of the diabetic foot once it has undergone partial amputation. To determine this, measures of healing, quality of life, and utilization costs associated with this approach will be analyzed. KCI believes that information obtained from this study will show V.A.C. NPWT can support efforts involving limb salvage of the diabetic foot, helping an effective, cost-efficient healthcare solution.

DETAILED DESCRIPTION:
Primary objective is to compare time required to achieve wound bed preparation between Subjects randomized to receive V.A.C. NPWT or MWT. Subjects with ALL the following are eligible for clinical trial enrollment:

Evidence of therapy controlled diabetes, as defined by the American Diabetes Association (ADA) of HbA1C less than or equal to 10%, within 90 days of screen or at time of screening, greater than or equal to 18 years of age, forefoot amputation less than or equal to 10 days old distal to the transmetatarsal level, not extending beyond the Lisfranc joint, receiving MWT allowed in the protocol for treatment of the study wound, Wound surface area measured as length x width of greater than or equal to 10 cm2, Subject is willing and able to provide written informed consent and comply with follow-up visit schedule and maintain a treatment diary, Adequate nutrition to enable wound healing as evidenced by a prealbumin level of greater than or equal to 16 mg/dl or an albumin level of greater than or equal to 3 g/dl within 7 days of screening or at the screening visit, Adequate perfusion in the affected extremity as evidenced by grade 1 or 2 PVR waveform as confirmed at screening, Non-pregnant female Subject of childbearing potential confirmed negative by serum HCG or surgically sterilized or unable to conceive.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of therapy controlled diabetes, as defined by the American Diabetes Association (ADA) of HgbA1C ≤10%, within 90 days of screening or at time of screening
* ≥18 years of age
* Forefoot amputation ≤ 8 days old distal to the transmetatarsal level, not extending beyond the Lisfranc's joint
* Receiving MWT allowed in the protocol for treatment of the study wound Protocol: V.A.C. 2006-19 Version 1.10 14 November 2007 Confidential/Proprietary Property of KCI, Inc. 28
* Wound surface area, measured as length x width, of ≥10 cm2
* Subject is willing and able to provide written informed consent, comply with follow-up visit schedule, and maintain a treatment diary
* Adequate nutrition to enable wound healing as evidenced by a pre-albumin level of

  ≥16 mg/dl or an albumin level of ≥3g/dl within 7 days of screening or at the screening visit
* Adequate perfusion in the affected extremity as evidenced by Grade 1 or 2 PVR waveform as confirmed at screening (see Section 7.1)
* Non-pregnant female Subject of child-bearing potential (confirmed negative by serum hCG), surgically sterilized, or unable to conceive

Exclusion Criteria:

* Untreated or refractory cellulitis of the wound with periwound erythema ≥3 cm
* Untreated or refractory osteomyelitis of the wound
* Untreated or refractory infection of the wound
* Exposed blood vessels in or around the wound
* Surgical revascularization of the affected extremity ≤10 days from study enrollment other than by percutaneous means
* Percutaneous revascularization of the affected extremity ≤2 days from study enrollment
* Grade 3-5 PVR waveforms
* Long-term (≥30 days) use of steroids (NOTE: Use of non-wound-indicated topical, optical or aerosol types of steroids are permitted at screening and throughout the clinical trial)
* Active Charcot disease of either lower extremity that will interfere with wound treatment
* Malignancy in the wound, around margins or any other malignancy requiring immunosuppressant therapy or chemotherapy
* Presence of necrotic tissue with eschar or slough that cannot be debrided
* Persistent periwound maceration of >96 hours
* Inadequate wound hemostasis that might impair wound healing
* Reported alcohol or drug abuse within the past 6 months
* Topical hypersensitivity or allergy to any disposable component of the V.A.C.® Protocol: V.A.C. 2006-19 Version 1.10 14 November 2007 Confidential/Proprietary Property of KCI, Inc. 29 NPWT System or to tape, dressings, or adhesives
* Female patients with plans to become pregnant during the study period
* Physical (i.e., venous sclerosis) or mental inability to undergo venipuncture for laboratory specimen collection
* Previous participation in this clinical study (VAC 2006-19)
* Participation in any other clinical study ≤30 days of enrollment
* Severe skin conditions (e.g. Meleney's ulcer, scleroderma) that may impair wound healing
* Connective tissue disease or collagen vascular disease (e.g. Ehlers-Danlos syndrome, systemic lupus erythematosus, rheumatoid arthritis) that may impair wound healing
* Hematological disorders or conditions (e.g. polycythemia vera, thrombocythemia, sickle-cell disease) that may impair wound healing
* History of clinically significant chronic anemia as evidenced by a hemoglobin concentration of <10.0 g/dL within ≤30 days of screening
* Severe venous insufficiency (with or without the presence of venous leg ulcers) that may impair wound healing
* Use of V.A.C.® NPWT System to the study wound ≤8 days prior to screening
* Use of any other suction device on the study wound within ≤8 days prior to screening
* Use of normothermic therapy (Warm-UP®) ≤8 days prior to screening
* Use of hyperbaric oxygen therapy (HBO) ≤30 days prior to screening
* Application of recombinant or autologous growth factors (e.g. Regranex® or Procuren®) on the study wound ≤8 days prior to screening
* Application of skin or dermal substitutes and dressings with living cells capable of producing growth factors (e.g. Oasis®, Apligraf®, Dermagraft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Blume, DPM, F.A.C.F.A.S, Principal Investigator — North American Center for Limb Preservation; Brent Bernstein, DPM, F.A.C.F.A.S, Principal Investigator — St. Lukes Allentown & Bethlehem; Marc Corriveau, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Vickie Driver, M.D., Principal Investigator — Boston University; Stephan Elkouri, MD, MSc, FRCSC, FAC, Principal Investigator — Centre Hospitalierde l'Universite' de Montreal (CHUM); Luis Esquerdo, DPM, Principal Investigator — Esquerdo Podiatric Center; Christopher Gauland, MD, Principal Investigator — Eastern Carolina Foot and Ankle; Vivian Halpern, MD, Principal Investigator — North Shore University Hospital; Jason Hanft, DPM, Study Director — Doctor's Research Network; Adam Landsman, DPM, PhD., Principal Investigator — Beth Israel Deaconess Medical Center Division of Podiatry, Baker 3; John Lantus, MD, Principal Investigator — St. Lukes-Roosevelt Hospital Center; James Mahoney, MD, FRCS, Principal Investigator — Division of Plastic Surgery- St. Michael's Hospital; Jose Mattei, MD, DPM, Principal Investigator — CTI Network Inc; Kenneth McIntyre, MD, Principal Investigator — Mike O'Callaghan Military Hospital; Christopher Moore, DPM, Principal Investigator — Moore Foot & Ankle Specialists, PA; Lili Moore, DPM, Principal Investigator — Moore Foot & Ankle Specialists, PA; Wyatt Payne, MD, Principal Investigator — Bay Pines VAHCS; Rodney Stuck, DPM, Principal Investigator — Hines VA Hospital; Jodi Walters, DPM, Principal Investigator — Southern Arizona VA Healthe Care System; Joseph Whitlark, MD, Principal Investigator — Comprehensive Wound Care, Inc; Thomas Zgonis, MD, Principal Investigator — University of Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | V.A.C. Therapy | Moist Wound Therapy (MWT)
Started | 10 | 9
Completed | 0 | 0
Not Completed | 10 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Not reported | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V.A.C. Therapy | Moist Wound Therapy (MWT) | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (13.15) | 55.9 (14.56) | 55.2 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 2
  White | 6 | 5 | 11
  Hispanic or Latino | 3 | 2 | 5
  Other: Arabic | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 2 | 0 | 2
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 100% Wound Closure
Time Frame: Day 84
Measure: Count of Participants; unit: Participants
Arm/Group | V.A.C. Therapy | Moist Wound Therapy (MWT)
Number analyzed (Participants) | 10 | 9
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 84
Description: Adverse Events were assessed at each protocol scheduled visit.
Arm/Group | V.A.C. Therapy | Moist Wound Therapy (MWT)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 5/10 | 3/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V.A.C. Therapy (N=10) | Moist Wound Therapy (MWT) (N=9)
Osteomyelitis (Infections and infestations) | 1 | 1
Patient fell at home, transported to ER by EMS (General disorders) | 0 | 1
Biliary pancreatitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Infected fracture hematoma (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Infected ulcer (Infections and infestations) | 1 | 0
Resuscitation (unknown diagnosis) (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days